CLINICAL TRIAL: NCT01596023
Title: Evaluation of Effect of Breathe Ventilation System on Work of Breathing in COPD Patients
Brief Title: Evaluation of Breathe NIOV System on Work of Breathing in Chronic Obstructive Lung Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Breathe Technologies, Inc. (Industry)
Collaborators: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: CP-00-0033
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Obstructive Lung Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIOV Ventilator (Experimental): Breathe NIOV Ventilator under various volume augmentation settings
  Interventions: Device: Breathe NIOV Ventilator

INTERVENTIONS:
Device: Breathe NIOV Ventilator — Portable, non invasive open ventilation system

SUMMARY:
The Breathe Ventilator is a lightweight, wearable ventilator that has received U.S. FDA clearance for use in patients with respiratory difficulty. The investigators believe that the Breathe NIOV system will reduce the work of the diaphragm and breathing by providing added tidal volume and oxygen. This will be a study in 14 patients with severe-to-very severe chronic obstructive lung disease (COPD) to assess their work of breathing while using the NIOV system as measured by esophageal and stomach pressures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is >18 years of age at time of consent.
2. Subject has diagnosis of severe COPD (GOLD stage III or IV) as demonstrated by a FEV1 < 50% predicted and FEV1/FVC ratio < 70% predicted.
3. Subject has increased inspiratory muscle work of breathing as evidenced by palpable sternocleidomastoid muscle contraction during inspiration

Exclusion Criteria:

1. Subject has acute exacerbation of COPD - within 1 week of acute hospitalization
2. Subject has respiratory rate at rest > 28/min
3. Subject requires > 5 L/min nasal O2/min to maintain O2sat > 90%
4. Subject has severe dyspnea at rest
5. Subject has swallowing disorders or chronic aspiration, prior esophageal surgery, or any other condition that would place the subject at risk during balloon placement.
6. Subject has history of pneumothorax secondary to lung bullae.
7. Subject is too cognitively impaired to give subjective ratings for visual analog scale
8. Subject has sensitivity or an allergy to lidocaine
9. Subject has known history of oxygen intolerance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pressure time product of the diaphragm (PTPdi) during use of the Breathe Ventilation System | 10 min
  Calculated using the area of the transdiaphragmatic pressure for the duration of inspiration

SECONDARY OUTCOMES:
Changes in PTP of the esophagus (PTPes), PTP per minute (PTPdi/min and PTPes/min | 10 Min
  Changes in PTP of the esophagus (PTPes), PTP per minute (PTPdi/min and PTPes/min)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hill, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States